CLINICAL TRIAL: NCT07263243
Title: Immediate Effect of Whole-Body Vibration on Cardiovascular Response and Functional Capacity in Overweight/Obese Young Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rokaia Ali Zainelabedeen Mohamed Toson, Assistant Professor of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 7699
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Overweight , Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Whole body vibration group) (Experimental): The study group (no = 13) underwent single session of whole-body vibration (WBV) of using the PowerPlate device.
  Interventions: Device: Whole-body vibration device
- Control group (Sham whole body vibration group) (Experimental): The sham WBV group (no=13) will stand on the same device with the vibtation shut off for single session.
  Interventions: Other: Sham whole body vibration

INTERVENTIONS:
Device: Whole-body vibration device — Whole-body vibration (WBV) training using the Power Plate Pro 7HC (Northbrook, USA). The vibration frequency was set at 30 Hz, with an amplitude of 2 mm.
  Arms: Study Group (Whole body vibration group)
Other: Sham whole body vibration — A sham Whole body vibration will be used . participants will stand on the device without actual vibrations.This control condition will be used to isolate the effects of WBV from other potential influences such as standing posture and time spent on the the platform.
  Arms: Control group (Sham whole body vibration group)

SUMMARY:
Obesity has become a major global public health issue, defined by an excessive accumulation of body fat that presents substantial health risks. Over 650 million adults worldwide suffer from obesity, which is defined as having a Body Mass Index (BMI) of 30 or higher. Obesity is becoming more common in both developed and developing countries. Sedentary lifestyles, unhealthy eating habits that include processed foods and sugars, and genetic factors are the main causes of the rising prevalence of obesity. Obesity is a multifactorial condition that affects physical appearance and self-esteem, while also having significant implications for long-term health, leading to decreased life expectancy and lower quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 to 25.
* normotensive (<140/90 mmHg).
* Their BMI was from 25 to 40 kg/m2.
* Sedentary (≤ 90min of regular exercise per week).

Exclusion Criteria:

* Having previously diagnosed with any chronic disease.
* Cardiorespiratory or neuromuscular conditions.
* Participating in any exercise program.
* Patients with a pacemaker.
* Pregnancy.
* Smoking.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 26 (Estimated)
Dates: Start 2026-01-24 (Estimated); Primary Completion 2026-02-24 (Estimated); Study Completion 2026-02-24 (Estimated)

PRIMARY OUTCOMES:
Brachial blood pressure | 1 day
  Systolic brachial blood pressure and diastolic brachial blood pressure will be measured using a blood pressure (BP) monitoring device after 15 minutes rest.
Heart rate | 1 day
  Heart rate will be measured using a pulse oximeter after 15 minutes rest.
Arterial O2 saturation | 1 day
  Arterial oxygen saturation of pulse oximetry (SpO2) were measured using a pulse oximeter.

SECONDARY OUTCOMES:
6-Minute walk test | 1 day
  The 6-Minute Walk Test (6MWT) is a simple, practical assessment used to measure functional exercise capacity. It evaluates how far a person can walk on a flat, hard surface (usually 30 meters) in six minutes. It is widely used in cardiology, pulmonology, and rehabilitation.
The Borg scale | 1 day
  The Borg Scale is a tool used to measure a person's perceived exertion and how hard they feel they are working during physical activity. It is commonly used during cardiac rehab, pulmonary rehab, exercise training, and clinical assessments. the scale ranges from 6 represents no exertion at all and to 20 represents maximal exertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Jouf University, Jouf, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes